CLINICAL TRIAL: NCT04784936
Title: Identification of Stroke at the Emergency Medical Dispatch Center
Acronym: IdStroke
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Katarina Bohm, PhD, Karolinska Institutet
Other Study IDs: Stroke2010/703-31/2
Record Dates: First submitted 2016-02-23; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A study to investigate how stroke is identified and whether FAST, face-arm-speech test, is used in the emergency medical dispatch centre in Stockholm. The study will also investigate when FAST is used, does it increase the identification of stroke? And if other factors can be identified as "markers" for more effective identification of stroke during the emergency call.

DETAILED DESCRIPTION:
Transcribed alarm calls are read through and analyzed using a qualitative method. Meaningful units are identified, coded and categorized. A phenomenological analysis is also applied to a separate analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who has called the emergency medical dispatch centre and also are diagnosed as stroke at Södersjukhuset during the study period.

Exclusion Criteria:

* Cases where needed documents and files are missing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who has called the emergency medical dispatch centre and also are diagnosed as stroke at Södersjukhuset during the study period.
Sampling Method: Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-10-30 (Actual)

PRIMARY OUTCOMES:
Frequency of stroke symptoms | 1 h
  A data collection tool assessing the frequency of stroke symptoms will be developed. The data collection tool will identify stroke symptoms presented by the caller during emergency calls and assess stroke symptoms in the Face-Arm-Speech-Time Test (FAST). Stroke symptoms will then be quantified into percentages for a descriptive analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Bohm, PhD, Principal Investigator — Karolinska Institutet, Intitution of clinical science and education, Södersjukhuset
Locations (1):
- Karolinska Institutet, Intitution of clinical science and education, Södersjukhuset, Stockholm, Sweden